CLINICAL TRIAL: NCT02752815
Title: Four Cycles of R-CHOP Followed by Four Cycles of Rituximab Versus Six Cycles of R-CHOP Followed by Two Cycles of Rituximab in the Treatment of de Novo, Low-risk, Non-bulky Diffuse Large B-cell Lymphoma.
Brief Title: Reduced Chemotherapy in Low Risk DLBCL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHL-006
Record Dates: First submitted 2016-04-20; First posted 2016-04-27 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Epirubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6R-CHOP+2R (Active Comparator): 6 cycles of R-CHOP Rituximab 375 mg/m2 IV d1 Cyclophosphamide 750mg/m2 IV d2 Epirubicin 70mg/m2 IV d2 Vincristine 1.4 mg/m2 IV d2 Prednisone 60 mg/m2 PO d2-6 Frequency 21days
  2 cycles of Rituximab monotherapy Rituximab 375 mg/m2 IV d1 Frequency 21days
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Epirubicin; Drug: Vincristine; Drug: Prednisone
- 4R-CHOP+4R (Experimental): 4 cycles of R-CHOP Rituximab 375 mg/m2 IV d1 Cyclophosphamide 750mg/m2 IV d2 Epirubicin 70mg/m2 IV d2 Vincristine 1.4 mg/m2 IV d2 Prednisone 60 mg/m2 PO d2-6 Frequency 21days
  2 cycles of Rituximab monotherapy Rituximab 375 mg/m2 IV d1 Frequency 21days
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Epirubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab
Drug: Cyclophosphamide
Drug: Epirubicin
Drug: Vincristine
Drug: Prednisone

SUMMARY:
This is a clinical trial to compare the efficacy and safety of four cycles of R-CHOP followed by four cycles of Rituximab with six cycles of R-CHOP followed by two cycles of Rituximab in the treatment of de novo, low-risk, non-bulky diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed de novo diffuse large B-cell lymphoma, complete response after 4 cycles of standard R-CHOP21
* Age>=14 y.o.,<=75 y.o.
* IPI=0-1
* non-bulky (largest diameter <7.5cm)
* ECOG =0-1
* Life expectancy>6 months
* Informed consented

Exclusion Criteria:

* Chemotherapy before
* Stem cell transplantation before
* History of malignancy, except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Uncontrollable cardio-cerebral vascular, coagulative, autoimmune, serious infectious disease
* Primary cutaneous, CNS DLBCL
* LVEF≤50%
* Other uncontrollable medical condition that may that may interfere the participation of the study
* Lab at enrollment(unless caused by lymphoma) Neutrophile<1.5*10^9/L Platelet<80*10^9/L Hemoglobulin<100g/L ALT or AST >2*ULN,AKP or bilirubin >1.5*ULN Creatinine>1.5*ULN
* Not able to comply to the protocol for mental or other unknown reasons
* Pregnant or lactation
* If HbsAg positive, should check HBV DNA, DNA positive patients cannot be enrolled. If HBsAg negative but HBcAb positive (whatever HBsAb status), should check HBV DNA,DNA positive patients cannot be enrolled.
* HIV infection

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2016-06-14 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2-year

SECONDARY OUTCOMES:
Overall survival | 2-year
Complete Response rate | 21 days after 8 cycles of treatment（each cycle is 21 days）
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Each cycle of treatment（each cycle is 21 days）and then every 3 months for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, MD, PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Shi Q, He Y, Yi HM, Mu RJ, Jiang XF, Fu D, Dong L, Qin W, Xu PP, Cheng S, Song Q, Chen SJ, Wang L, Zhao WL. Positron emission tomography-adapted therapy in low-risk diffuse large B-cell lymphoma: results of a randomized, phase III, non-inferiority trial. Cancer Commun (Lond). 2023 Aug;43(8):896-908. doi: 10.1002/cac2.12462. Epub 2023 Jul 4. PMID 37403255